CLINICAL TRIAL: NCT00233805
Title: A Randomized Study With the Sirolimus Coated Modified BX Velocity Balloon-Expandable Stent in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: The Initial Double-Blind Drug-Eluting Stent vs Bare-Metal Stent Study.
Acronym: RAVEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Director Clinical Affairs, Cordis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC00-01
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bare metal Bx Velocity™ Balloon-Expandable Stent mounted on the Raptor® rapid exchange delivery system
  Interventions: Device: Bare metal Bx Velocity™
- 2 (Experimental): Sirolimus coated modified Bx Velocity™ Balloon-Expandable Stent mounted on the Raptor® rapid exchange delivery system
  Interventions: Device: Sirolimus coated Bx Velocity™

INTERVENTIONS:
Device: Sirolimus coated Bx Velocity™ — drug-eluting stent
  Arms: 2
Device: Bare metal Bx Velocity™ — bare-metal stent
  Arms: 1

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the sirolimus coated Bx VELOCITY stent in reducing angiographic in-stent late loss in de novo native coronary lesions as compared to the bare metal Bx VELOCITY balloon-expandable stent. Both stents will be mounted on the Raptor Rapid Exchange Delivery Stent System.

DETAILED DESCRIPTION:
This is a multicenter (19 sites), prospective, randomized study. This study has a 2 arm design assessing the safety and effectiveness of the sirolimus coated BxTM VELOCITY stent to the bare metal BxTM VELOCITY stent, both mounted on the Raptorâ Rapid Exchange Stent Delivery System. A total of 220 patients will be entered in the study and will be randomized on a 1:1 basis. Patients will be randomized to the coated or uncoated BX VELOCITY stent. Therefore, neither the Investigator nor the patient will know which stent will be implanted. Patients will be followed for twelve months post-procedure, with all patients having a repeat angiography at 6 months. An ancillary study with in-stent IVUS measurements at 6 months follow-up will be performed in all patients of 6 pre-selected clinical sites. It is assumed that these sites will enroll more than 90 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
2. Single treatment of de novo lesion in a coronary artery which can be appropriately covered by a study stent of 18mm in length in patients with single or multivessel disease; patients with multiple lesions can be included only if the other lesions do not require treatment;
3. Target lesion is >= 2.5 and <= 3.5mm in diameter (visual estimate);
4. Target lesion is located in a native coronary artery which can be covered by one stent (single lesion);
5. Target lesion stenosis is >50% and <100% (TIMI I) (visual estimate).

Exclusion Criteria:

1. A Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal;
2. Unprotected left main coronary disease with >=50% stenosis;
3. Have an ostial target lesion;
4. Angiographic evidence of thrombus within target lesion;
5. Calcified lesions which cannot be successfully predilated;
6. Ejection fraction <=30%;
7. Totally occluded vessel (TIMI 0 level);
8. Target lesion involves bifurcation including a side branch >=2.5mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require side branch stenting which is likely to occur if side branch is diseased and intended to be stented;
9. Planned Direct Stenting.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2000-08; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Angiographic in-stent late loss as determined by Quantitative Coronary Angiography. | 6 months follow-up

SECONDARY OUTCOMES:
In-stent mean %DS by QCA | post-procedure
In-target vessel segment MLD | 6 months
In-stent MLD | 6 months
Target Lesion Revascularization | 6 and 12 months; or 2, 3, 4 and 5 years
Target Vessel Revascularization | 6 and 12 months; or 2, 3, 4 and 5 years
Major Adverse Cardiac Events | 30 days; 6 and 12 months; or 2, 3, 4 and 5 years;
Neo-intimal growth assessed by IVUS | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Morice, MD, Principal Investigator — Institut Hospitalier Jacques Cartier
Locations (1):
- Dr Marie-Claude Morice, Massy, France

REFERENCES:
- [Background] Hoffmann R, Morice MC, Moses JW, Fitzgerald PJ, Mauri L, Breithardt G, Schofer J, Serruys PW, Stoll HP, Leon MB. Impact of late incomplete stent apposition after sirolimus-eluting stent implantation on 4-year clinical events: intravascular ultrasound analysis from the multicentre, randomised, RAVEL, E-SIRIUS and SIRIUS trials. Heart. 2008 Mar;94(3):322-8. doi: 10.1136/hrt.2007.120154. Epub 2007 Aug 29. PMID 17761505
- [Result] Fajadet J, Morice MC, Bode C, Barragan P, Serruys PW, Wijns W, Constantini CR, Guermonprez JL, Eltchaninoff H, Blanchard D, Bartorelli A, Laarman GJ, Perin M, Sousa JE, Schuler G, Molnar F, Guagliumi G, Colombo A, Ban Hayashi E, Wulfert E. Maintenance of long-term clinical benefit with sirolimus-eluting coronary stents: three-year results of the RAVEL trial. Circulation. 2005 Mar 1;111(8):1040-4. doi: 10.1161/01.CIR.0000156334.24955.B2. Epub 2005 Feb 21. PMID 15723977
- [Result] Abizaid A, Costa MA, Blanchard D, Albertal M, Eltchaninoff H, Guagliumi G, Geert-Jan L, Abizaid AS, Sousa AG, Wuelfert E, Wietze L, Sousa JE, Serruys PW, Morice MC; Ravel Investigators. Sirolimus-eluting stents inhibit neointimal hyperplasia in diabetic patients. Insights from the RAVEL Trial. Eur Heart J. 2004 Jan;25(2):107-12. doi: 10.1016/j.ehj.2003.11.002. PMID 14720526
- [Result] Regar E, Serruys PW, Bode C, Holubarsch C, Guermonprez JL, Wijns W, Bartorelli A, Constantini C, Degertekin M, Tanabe K, Disco C, Wuelfert E, Morice MC; RAVEL Study Group. Angiographic findings of the multicenter Randomized Study With the Sirolimus-Eluting Bx Velocity Balloon-Expandable Stent (RAVEL): sirolimus-eluting stents inhibit restenosis irrespective of the vessel size. Circulation. 2002 Oct 8;106(15):1949-56. doi: 10.1161/01.cir.0000034045.36219.12. PMID 12370218
- [Result] Serruys PW, Degertekin M, Tanabe K, Abizaid A, Sousa JE, Colombo A, Guagliumi G, Wijns W, Lindeboom WK, Ligthart J, de Feyter PJ, Morice MC; RAVEL Study Group. Intravascular ultrasound findings in the multicenter, randomized, double-blind RAVEL (RAndomized study with the sirolimus-eluting VElocity balloon-expandable stent in the treatment of patients with de novo native coronary artery Lesions) trial. Circulation. 2002 Aug 13;106(7):798-803. doi: 10.1161/01.cir.0000025585.63486.59. PMID 12176950
- [Result] Morice MC, Serruys PW, Barragan P, Bode C, Van Es GA, Stoll HP, Snead D, Mauri L, Cutlip DE, Sousa E. Long-term clinical outcomes with sirolimus-eluting coronary stents: five-year results of the RAVEL trial. J Am Coll Cardiol. 2007 Oct 2;50(14):1299-304. doi: 10.1016/j.jacc.2007.06.029. Epub 2007 Sep 17. PMID 17903626
- [Derived] Spaulding C, Daemen J, Boersma E, Cutlip DE, Serruys PW. A pooled analysis of data comparing sirolimus-eluting stents with bare-metal stents. N Engl J Med. 2007 Mar 8;356(10):989-97. doi: 10.1056/NEJMoa066633. Epub 2007 Feb 12. PMID 17296825